CLINICAL TRIAL: NCT06115096
Title: Exploration of Intracardiac Geometry and Hemodynamics During HeartMate 3 Therapy: A Novel Approach Using Photon-Counting CT and Computational Fluid Dynamics
Brief Title: Cardiac Hemodynamics During Left Ventricular Assist
Acronym: FlowVAD
Status: Recruiting | Type: Observational
Sponsor: Region Östergötland (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Hans Granfeldt, Senior consultant, cardiothoracic surgery (MD/PhD), deputy operational manager, Region Östergötland
Other Study IDs: FlowVAD
Record Dates: First submitted 2023-10-16; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
Keywords: Left ventricular assist device (LVAD); Computed tomography (CT); Photon-counting Computed tomography (PCCT); Hemodynamics; Computational fluid dynamics (CFD)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to exploratively investigate intracardiac geometry and hemodynamics in patients with ongoing HeartMate 3-therapy in the Swedish Southeast Healthcare region. The main question it aims to answer is:

- How do different flow levels in the HeartMate 3 left ventricular assist system influence intracardiac geometry and hemodynamics?

Participating research subjects are called upon to undergo three followed photon-counting CT scans, as well as certain echocardiographic imaging, all in one session. The research subject's HeartMate device is connected to software that allows for variations in the pump's flow between these image collections. Analyzed variables includes three-dimensional geometry, CFD-computed parameters such as blood velocity, pressure, turbulence, and blood stasis. The variables are related with device settings and, alongside, selected echocardiographic measurements and patient details such as age, BMI, and diagnostic codes for both method validation and comprehensive perspective.

DETAILED DESCRIPTION:
1. BACKGROUND

   In recent years, the use of the mechanical circulatory support device, HeartMate 3 (HM3) (Abbott Laboratories, Lake Forest, IL), has garnered significant attention in the realm of circulatory support for advanced heart failure. The tangible advantages of the HM3, including enhanced hemocompatibility leading to reduced thromboembolic events and improved survival rates compared to its predecessors. The transition towards HM3 is particularly noteworthy as the system is not only likely to serve as a bridge to heart transplantation or decision-making but is increasingly being discussed as an effective destination therapy. Despite these advancements, there remains an imperative for meticulous hemodynamic monitoring throughout any mechanical circulatory support treatment. Traditionally, echocardiography has been predominantly employed as the hemodynamic imaging modality. However, echocardiographic evaluations of these patients present notable challenges, especially concerning shadows from the pump's metal, making it difficult to fully comprehend cardiac function and hemodynamics during the treatment.

   Over the past decade, computed tomography (CT) has seen rapid advancements, with modern equipment now facilitating high-resolution anatomical imaging of the heart throughout the cardiac cycle (4D CT). Until recently, however, CT also posed a challenge for the examination of patients with mechanical circulatory support devices due to significant metal artifacts. The newly introduced photon-counting computed tomography (PC-CT), however, now enables scans that yield higher resolution images with reduced metal artifacts. From time-resolved CT, functional information can subsequently be derived and extracted. Techniques for automatic tracking of cardiac wall motion throughout the cardiac cycle, along with the utilization of computational dynamics to numerically solve fluid mechanical equations have previously been shown, which have proven to enable simulations of intracardiac hemodynamic maps.

   The increasing indications for treatment with mechanical circulatory support underscore the current demand for continuously improved care quality and clinical understanding of this therapeutic option. Although the treatment enhances both prognosis and quality of life, serious and fatal complications remain recurrent. To the knowledge of the investigators, there has yet been no conducted research addressing the potential application of the novel PC-CT in patients with mechanical circulatory support devices, and certainly none that have established numerical frameworks on this data in an attempt to compute, visualize, and exploratively understand intracardiac hemodynamics during the treatment.

   1.2 OBJECTIVES

   1.2.1 AIM

   The aim of this observational study is to exploratively investigate intracardiac geometry and hemodynamics in patients with ongoing HeartMate 3-therapy in the Swedish Southeast Healthcare region.

   1.2.2 PRIMARY SCIENTIFIC QUESTION

   How do different flow levels in the HeartMate 3 left ventricular assist device influence intracardiac geometry and hemodynamics?
2. METHODS

2.1 STUDY DESIGN

This study has an explorative analytic (multiple) cross-sectional design. The study seeks to uncover new insights, patterns, and associations within the data, partly without predetermined hypotheses. Further, the study investigates relationships or associations between variables to derive meaningful conclusions from the data. The study will examine three distinct observations of the variables, wherein the subjects' device settings will vary. These observations, however, will be executed in close temporal proximity, with intervals of approximately 15 minutes between each. As such, while the study does not fully conform to the criteria of a multiple cross-sectional study design, it also does not align with a traditional one-time-point cross-sectional approach.

2.2 OVERALL SETTING

Participating research subjects are called upon to undergo three followed PC-CT scans, as well as certain echocardiographic imaging, all in one session. The research subject's HM3 is connected to software that allows for variations in the pump's flow between these image collections. All examinations will be performed at Center for Medical Image Science and Visualization (CMIV) at Linköping University, Sweden. Recruitment and examination within the study will undergo during January-December 2023. The study has been approved by the Swedish ethics review authority (Reference number: 2022-06934-01).

2.2 PARTICIPANTS

All patients within the Swedish Southeastern healthcare region, encompassing Östergötland, Jönköping, and Kalmar counties, who meet the inclusion criteria and none of the exclusion criteria, will be invited to participate in this study during 2023. Screening for inclusion is conducted by the LVAD-responsible physicians within the Cardiology Department at Linköping University Hospital.

2.3 VARIABLES

Regarding specification of variables that will be studied, it is essential to clarify that due to the exploratory nature of the research and the intricate dynamics inherent to both using numerical frameworks for calculating intracardiac hemodynamic maps and the dynamic geometric nature of time-resolved CT, all variables at the study onset are not pre-defined. As the analysis progresses, and the full depth of the data becomes apparent, additional variables may be identified and incorporated. Subsequent decision-making process relating to the inclusion or exclusion of these newly discovered variables will be rigorously documented to ensure transparency and robustness in the study approach.

Quantified variables will be compared with respect to the pump's estimated flow (L/min), power (W), pulsatility index, and rotor speed (rpm). Whenever possible, based on image quality, the results will also be related to and compared with echocardiographic measurements to discuss the validity of the method. To reduce the risk of unintended confounding factors and to minimize the potential for bias, several baseline data regarding the included research subjects will also be collected. These variables include age (years), gender, HM3 implantation date body mass index (BMI, kg/m^2), and cardiovascular diagnostic codes (ICD-10), blood count (cells/μL or x10^9/L), electrolytes (mmol/L), liver function tests (U/L or µkat/L for enzymes, and g/dL or µmol/L for substances), lactate dehydrogenase (U/L), NT-proBNP (pg/mL or ng/L), and procalcitonin (ng/mL).

2.4 DATA SOURCES AND MEASUREMENTS

2.4.1 PC-CT EXAMINATION PCCT-examinations will be performed utilizing a CE-marked photon-counting computed tomography system (NAETOM Alpha, Siemens Healthineer, Erlangen, Germany). The acquisitions will be effectuated at 120 kVp with image quality (IQ) levels set at 70. A biphasic contrast administration protocol will be employed to guarantee opacification across all four cardiac chambers. The entirety of the scan range will undergo multiphase reconstructions at intervals corresponding to every 5% of the cardiac cycle, culminating in 20 distinct phases. Acquired CT-images were relayed to the institution's Picture Archiving and Communication System (PACS, IDS7, Sectra Medical Systems, Linköping, Sweden).

2.4.2 SEGMENTATION AND WALL MOTION TRACKING

The motion of the endocardium will be tracked from the acquired CT-data. In this process, the endocardium will semi-automatically be outlined with ITK-SNAP (version 3.8.0). The geometry will then be refined using Ansys SpaceClaim version 2019 R3 (Ansys Inc, Canonsburg, PA 15317 USA). Following this, the endocardial surface will be reshaped using a non-rigid iterative closed point method to align with threshold-based segmentations from the remaining 19 cardiac phases.

2.4.3 CFD SIMULATIONS

Blood flow velocity, absolute pressure, turbulence kinetic energy and blood stasis and other potential hemodynamic variables will be derived using Computational Fluid Dynamics (CFD) simulations, considering the participant-specific cardiac wall motion. The CFD simulations will be performed using Ansys Fluent version 2019 R3, based on the process previously validated using 4D flow MRI. Two cardiac models will be applied. The left model will include pulmonary veins, left atrium, left ventricle, the HM3, outflow graft, left ventricular outflow tract and ascending aorta. The right model will include superior vena cava, inferior vena cava, right atrium, right ventricle, right ventricular outflow tract and the pulmonary artery. All openings will be modelled as pressure openings, with the flow rate resulting from the motion of the endocardium.

2.4.3 PUMP VARIABLES AND BLOOD PRESSURE

Prior to every individual CT-scan, estimated flow (L/min), power (W), pulsatility index, and rotor speed (rpm), will be acquired from the HeartMate 3 System Monitor together with systolic blood pressure (mmHg), acquired using doppler technology of the radial artery. These details will be transferred to an established dataset within the project.

2.4.5 ECHOCARDIOGRAPHY

Selected echocardiographic imaging will be conducted between each CT scan. The specified protocol for the study is derived from the routine clinical protocol used to examine this patient group but is selected based on the time aspect of the full examination in the research project. Clinical staff experienced in these examinations will perform the tests.

2.4.6 PATIENT CHARACTERISTICS

Characteristic variables of the research subjects will be obtained from the medical record of the research subjects. Furthermore, results from the most recent clinical blood tests will be obtained. These details will be transferred to an established dataset within the project.

2.5 BIAS

Due to the exploratory nature of the study, there are inherent risks of both systematic and non-systematic bias. Firstly, the variables to be studied are not entirely predefined at the outset due to the research's exploratory design, which may introduce bias. To counteract this, the decision-making process surrounding the inclusion or exclusion of emergent variables will be meticulously documented to ensure transparency and robustness in the research methodology. Another significant consideration in this study is the use of CFD simulations. These simulations, while powerful in modeling fluid dynamics within the cardiovascular system, are susceptible to biases based on the input parameters, boundary conditions, and numerical methods employed. The chosen mesh resolution, turbulence models, and assumptions about blood rheology can all influence the results. To bolster the validity of the quantified CFD results, a key validation attempt in this study is the inclusion of echocardiography assessments. However, the echocardiographic image quality will vary between patients, which in itself can introduce bias and impair the possibilities for adequate validation of the CFD simulations.

2.6 STUDY SIZE

Determining the requisite sample size for this project is a challenge due to the method not having been previously evaluated. Given this context, the investigators have thus drawn upon the available literature from echocardiography studies and attempted to derive clinically significant differences based on pump settings from this. The study aims to recruit up to 35 participants to ensure interpretable results.

2.7 STATISTICAL METHODS

Inter-group comparisons will be performed using two-sample t-test. To assess the association between variables, such as CFD-variables and geometrical parameters, linear regression analysis will be performed. All statistical computations will be done using MATLAB R2021b and the significance level will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Connected to Linköping University Hospital ((situated in the Swedish Southeastern healthcare region)
* Treatment with HeartMate 3 and implanted for > 6 months ago
* Age >18 years.

Exclusion Criteria:

* Reduced kidney function (eGFR below 45 ml/min/1.73m2).
* Known iodine contrast allergy
* In case of untreated manifest hyperthyroidism
* In case of suspected/newly diagnosed thyroid cancer where radioiodine examination/treatment may be relevant
* Myasthenia Gravis
* Ongoing pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HeartMate 3 patients within the Swedish Southeastern healthcare region, encompassing Östergötland, Jönköping, and Kalmar counties, who meet the inclusion criteria and none of the exclusion criteria, will be invited to participate in this study during 2023. Screening for inclusion is conducted by the LVAD-responsible physicians within the Cardiology Department at Linköping University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic Variables | Observations are made at a single point in time. No follow-up of outcomes are analyzed. Post-processing and analysis of both hemodynamic and geometric data are performed through study completion, an average of 1 year.
  Intracardiac hemodynamic variables such as blood flow velocity maps (m/s), absolute pressure maps (mmHg), turbulence kinetic energy maps (TKE), and blood stasis maps will be calculated both intracardiac and in the pump's outflow graft.
  It is essential to clarify that due to the exploratory nature of the research and the intricate dynamics inherent to both using numerical frameworks for calculating intracardiac hemodynamic maps and the dynamic geometric nature of time-resolved CT, all variables at the study onset are not pre-defined. As the analysis progresses, and the full depth of the data becomes apparent, additional variables may be identified and incorporated. Subsequent decision-making process relating to the inclusion or exclusion of these newly discovered variables will be rigorously documented to ensure transparency and robustness in the study approach.
Intracardiac Geometry | Observations are made at a single point in time. No follow-up of outcomes are analyzed. Post-processing and analysis of both hemodynamic and geometric data are performed through study completion, an average of 1 year.
  Intracardiac volumes (ml) will be calculated for the left atrium, left ventricle, right ventricle and right atrium over the cardiac cycle (20 phases).
  It is essential to clarify that due to the exploratory nature of the research and the intricate dynamics inherent to both using numerical frameworks for calculating intracardiac hemodynamic maps and the dynamic geometric nature of time-resolved CT, all variables at the study onset are not pre-defined. As the analysis progresses, and the full depth of the data becomes apparent, additional variables may be identified and incorporated. Subsequent decision-making process relating to the inclusion or exclusion of these newly discovered variables will be rigorously documented to ensure transparency and robustness in the study approach.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Granfeldt, MD/PhD, Principal Investigator — Region Östergötland
Locations (1):
- Linköping University Hospital, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldstein DJ, Naka Y, Horstmanshof D, Ravichandran AK, Schroder J, Ransom J, Itoh A, Uriel N, Cleveland JC Jr, Raval NY, Cogswell R, Suarez EE, Lowes BD, Kim G, Bonde P, Sheikh FH, Sood P, Farrar DJ, Mehra MR. Association of Clinical Outcomes With Left Ventricular Assist Device Use by Bridge to Transplant or Destination Therapy Intent: The Multicenter Study of MagLev Technology in Patients Undergoing Mechanical Circulatory Support Therapy With HeartMate 3 (MOMENTUM 3) Randomized Clinical Trial. JAMA Cardiol. 2020 Apr 1;5(4):411-419. doi: 10.1001/jamacardio.2019.5323. PMID 31939996
- [Background] Gupta V, Lantz J, Henriksson L, Engvall J, Karlsson M, Persson A, Ebbers T. Automated three-dimensional tracking of the left ventricular myocardium in time-resolved and dose-modulated cardiac CT images using deformable image registration. J Cardiovasc Comput Tomogr. 2018 Mar-Apr;12(2):139-148. doi: 10.1016/j.jcct.2018.01.005. PMID 29402736
- [Background] Imamura T, Chung B, Nguyen A, Sayer G, Uriel N. Clinical implications of hemodynamic assessment during left ventricular assist device therapy. J Cardiol. 2018 Apr;71(4):352-358. doi: 10.1016/j.jjcc.2017.12.001. Epub 2017 Dec 26. PMID 29287808
- [Background] Imamura T, Jeevanandam V, Kim G, Raikhelkar J, Sarswat N, Kalantari S, Smith B, Rodgers D, Besser S, Chung B, Nguyen A, Narang N, Ota T, Song T, Juricek C, Mehra M, Costanzo MR, Jorde UP, Burkhoff D, Sayer G, Uriel N. Optimal Hemodynamics During Left Ventricular Assist Device Support Are Associated With Reduced Readmission Rates. Circ Heart Fail. 2019 Feb;12(2):e005094. doi: 10.1161/CIRCHEARTFAILURE.118.005094. PMID 30704291
- [Background] Lantz J, Gupta V, Henriksson L, Karlsson M, Persson A, Carlhall CJ, Ebbers T. Intracardiac Flow at 4D CT: Comparison with 4D Flow MRI. Radiology. 2018 Oct;289(1):51-58. doi: 10.1148/radiol.2018173017. Epub 2018 Jun 26. PMID 29944089
- [Background] Lantz J, Henriksson L, Persson A, Karlsson M, Ebbers T. Patient-Specific Simulation of Cardiac Blood Flow From High-Resolution Computed Tomography. J Biomech Eng. 2016 Dec 1;138(12). doi: 10.1115/1.4034652. PMID 27618494
- [Background] Mehra MR, Naka Y, Uriel N, Goldstein DJ, Cleveland JC Jr, Colombo PC, Walsh MN, Milano CA, Patel CB, Jorde UP, Pagani FD, Aaronson KD, Dean DA, McCants K, Itoh A, Ewald GA, Horstmanshof D, Long JW, Salerno C; MOMENTUM 3 Investigators. A Fully Magnetically Levitated Circulatory Pump for Advanced Heart Failure. N Engl J Med. 2017 Feb 2;376(5):440-450. doi: 10.1056/NEJMoa1610426. Epub 2016 Nov 16. PMID 27959709
- [Background] Mehra MR, Uriel N, Naka Y, Cleveland JC Jr, Yuzefpolskaya M, Salerno CT, Walsh MN, Milano CA, Patel CB, Hutchins SW, Ransom J, Ewald GA, Itoh A, Raval NY, Silvestry SC, Cogswell R, John R, Bhimaraj A, Bruckner BA, Lowes BD, Um JY, Jeevanandam V, Sayer G, Mangi AA, Molina EJ, Sheikh F, Aaronson K, Pagani FD, Cotts WG, Tatooles AJ, Babu A, Chomsky D, Katz JN, Tessmann PB, Dean D, Krishnamoorthy A, Chuang J, Topuria I, Sood P, Goldstein DJ; MOMENTUM 3 Investigators. A Fully Magnetically Levitated Left Ventricular Assist Device - Final Report. N Engl J Med. 2019 Apr 25;380(17):1618-1627. doi: 10.1056/NEJMoa1900486. Epub 2019 Mar 17. PMID 30883052
- [Background] Ohlsson L, Moreira ADL, Back S, Lantz J, Carlhall CJ, Persson A, Hedman K, Chew MS, Dahlstrom N, Ebbers T. Enhancing students' understanding of cardiac physiology by using 4D visualization. Clin Anat. 2023 Apr;36(3):542-549. doi: 10.1002/ca.24009. Epub 2023 Feb 6. PMID 36695446
- [Background] Rosenbaum AN, Geske JB, Stulak JM, Kushwaha SS, Clavell AL, Behfar A. Left Ventricular Hemodynamics and Relationship With Myocardial Recovery and Optimization in Patients Supported on CF-LVAD Therapy. J Card Fail. 2022 May;28(5):799-806. doi: 10.1016/j.cardfail.2021.12.008. Epub 2021 Dec 17. PMID 34929296
- [Background] Stainback RF, Estep JD, Agler DA, Birks EJ, Bremer M, Hung J, Kirkpatrick JN, Rogers JG, Shah NR; American Society of Echocardiography. Echocardiography in the Management of Patients with Left Ventricular Assist Devices: Recommendations from the American Society of Echocardiography. J Am Soc Echocardiogr. 2015 Aug;28(8):853-909. doi: 10.1016/j.echo.2015.05.008. No abstract available. PMID 26239899
- [Background] Uriel N, Colombo PC, Cleveland JC, Long JW, Salerno C, Goldstein DJ, Patel CB, Ewald GA, Tatooles AJ, Silvestry SC, John R, Caldeira C, Jeevanandam V, Boyle AJ, Sundareswaran KS, Sood P, Mehra MR. Hemocompatibility-Related Outcomes in the MOMENTUM 3 Trial at 6 Months: A Randomized Controlled Study of a Fully Magnetically Levitated Pump in Advanced Heart Failure. Circulation. 2017 May 23;135(21):2003-2012. doi: 10.1161/CIRCULATIONAHA.117.028303. Epub 2017 Apr 6. PMID 28385948
- [Background] Zhou W, Bartlett DJ, Diehn FE, Glazebrook KN, Kotsenas AL, Carter RE, Fletcher JG, McCollough CH, Leng S. Reduction of Metal Artifacts and Improvement in Dose Efficiency Using Photon-Counting Detector Computed Tomography and Tin Filtration. Invest Radiol. 2019 Apr;54(4):204-211. doi: 10.1097/RLI.0000000000000535. PMID 30562270